CLINICAL TRIAL: NCT01593995
Title: Phase II Trial of Epidermal Growth Factor Ointment for Patients With Erlotinib Related Skin Effects
Brief Title: EGF Ointment for Erlotinib Skin Lesion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, Sung Yong Oh, Department of Internal Medicine, Dong-A University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAU-12-01(ML25441)
Record Dates: First submitted 2012-05-05; First posted 2012-05-08 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Non-small Cell Lung Cancer; Pancreatic Cancer
Keywords: Erlotinib; Skin side effect; EGF ointment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms | interventions — Epidermal Growth Factor; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EGF ointment (Experimental)
  Interventions: Drug: Epidermal growth factor (EGF) ointment

INTERVENTIONS:
Drug: Epidermal growth factor (EGF) ointment — EGF Ointment evenly apply to skin lesion every 12 hr/ day. If the skin lesion has been no improvement even though EGF ointment applied for 8 weeks, stopped study and assess it as "no effect"
  Other Names: Sesal Yeongo

SUMMARY:
Epidermal growth factor receptor-tyrosin kinase inhibitor (EGFR-TKI, Erlotinib) has demonstrated its efficacy in patients with non-small cell lung cancer and pancreatic cancer. But, their use is associated with dermatologic reactions of varying severity. Incidence of Erlotinib related skin effect (ERSE) was reported ~75% in NSCLC and pancreatic cancer phase III trials. Even though the dermatologic reactions could be a surrogated marker, it may be cause of dose modification. Also, it could give significant physical and psycho-social discomfort to patients. However, there is still a wide variety of drugs used- including, steroid, antibiotics, and vitamin D without any clear evidence based management recommendation.

The role of epidermal growth factor (EGF) has been extensively investigated in normal and pathological wound healing. It is implicated in keratinocyte migration, fibroblast function and the formation of granulation tissue. The first growth factor to be isolated growth factor therapy has progressed into clinical practice in the treatment of wounds.

Therefore, the investigators propose an epidermal growth factor ointment apply for patients with Erlotinib related skin effects.

DETAILED DESCRIPTION:
Erlotinib

Advances in the knowledge of tumor biology and mechanisms of oncogenesis has granted the singling out of several molecular targets for NSCLC treatment. Among these targets, epidermal growth factor receptor (EGFR), or HER1, has received particular attention in lung cancer treatment. EGFR is a transmembrane receptor found primarily on cells of epithelial origin. Autophosphorylation of its intracellular domain initiates a cascade of events leading to cell proliferation. EGFR is commonly expressed at a high level in a variety of solid tumors and it has been implicated in the control of cell survival, proliferation, metastasis and angiogenesis. The main pharmacological strategies in clinical development for therapeutic inhibition of EGFR are monoclonal antibodies to antagonize ligand-receptor binding, and small-molecules to inhibit tyrosine kinase domain activation. The main EGFR inhibitors are cetuximab, an anti-EGFR monoclonal antibody, and Erlotinib an EGFRtyrosine kinase inhibitor. The key indications for clinical use are colorectal cancer and head and neck cancer for cetuximab and NSCLC for Erlotinib. Erlotinib, a quinazolin-4-amine, is a highly potent, orally available, reversible inhibitor of EGFR tyrosine kinase. Erlotinib, in a phase III randomized placebo-controlled trial, has been proven to prolong survival (6.7 months versus 4.7 months for Erlotinib and for placebo respectively, p = 0.001) in NSCLC patients after first or second line chemotherapy. The analysis of quality of life and time to deterioration of patients reported symptoms showed statistically and clinically meaningful benefit for patients randomized to Erlotinib. Moreover, Erlotinib resulted active (response rate of 8.9%) and safe (only 5% of patients discontinued treatment for toxicity). Following this trial, Erlotinib has been approved by Food and Drug Administration and Committee for Medicinal Products for Human use in chemotherapy-pretreated advanced NSCLC. Skin rash is a common side-effect of all HER1/EGFR inhibitors.

EGF ointment

Rash affecting the skin above the waist, is the most common adverse event associated with Erlotinib, and generally develops within 7-10 days of starting treatment. Skin rash may spontaneously resolve and reappear and it is reversible following drug discontinuation. However, when it develops, this chronic side-effect is very distressing for the patient. The increasing use of EGFR-targeted agents and specifically of Erlotinib in NSCLC treatment, and simultaneously the lack of clinical trials on this topic, makes rash management and etiology investigation high priorities.

It has been reported that repeated treatment with EGF increases the epithelial cell proliferation in a dose dependent manner and accelerates the wound healing process, whereas a single EGF treatment has no noticeable effect on the wound-healing rate. There have been many studies aimed at developing a topical formulation with the sustained and stable pharmacological properties of recombinant human EGF (rhEGF). And the rh-EGF concentration between 1 and 5 ug/g can be seen as the ideal concentration to achieve the most efficient results for acute wounds with partial thickness defects.

ELIGIBILITY:
Inclusion Criteria:

* Age :older than 20
* ECOG performance status 0 -2
* Histologically lung cancer or Pancreatic Cancer
* Patients take Erlotinib following the reason Clinical failure of the prior therapy locally advanced or metastatic NSCLC The 1ST line using in combination with Gemcitabine for locally advanced, unresectable or metastatic Pancreatic Cancer(Adenocarcinoma)
* Patients who have Erlotinib-treatment related skin lesions Gr≥2 (NCI-CTC V3.0).
* A patient with at least one measurable primary lesion of which the diameter is confirmed to be 10mm in Spiral CT or multidetector CT (MD CT), or 20 mm or longer in conventional CT (it should be used by a consistent method during the study period).
* The following laboratory test results:

Creatinine clearance ≥ 60ml/min Number of absolute neutrophil counts (ANC) > 1.5 x 109/L Number of thrombocytes > 100 x 109/L Total bilirubin < 2x upper limit of normal ALAT, ASAT < 3 x upper limit of normal (in case of liver metastasis, 5 x upper limit of normal) Alkaline phosphatase < 3 x upper limit of normal (in case of liver metastasis, 5 x upper limit of normal)

* A patient with the willingness to comply with the study protocol during the study period and capable of complying with it.
* A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

* A patient with previous active or passive immunotherapy.
* A pregnant or lactating patient
* A patient of childbearing potential without being tested for pregnancy at baseline for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential.)
* A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications.
* A patient with history of dermatologic care (except transient urticaria) within 4 weeks
* A patient with clinically significant (i.e. active) heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmias, etc) or myocardial infarction within past 12 months.
* A patient with interstitial pneumonia or diffused symptomatic fibrosis of the lungs.
* Organ allogenic transplantation requiring immunosuppressive therapy. Any waiver of these inclusion and exclusion criteria must be approved by the investigator and the sponsor on a case-by case basis prior to enrolling the subject.
* Known allergies, hypersensitivity, or intolerance to Study drugs, Chemotherapy drugs using this Clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Improvement of skin lesion grading by NCI-CTC v3.0 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Oh, M.D.,Ph.D., Study Director — Onclogy Division, Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Busan, South Korea

REFERENCES:
- [Derived] Hwang IG, Kang JH, Oh SY, Lee S, Kim SH, Song KH, Son C, Park MJ, Kang MH, Kim HG, Lee J, Park YS, Sun JM, Kim HJ, Kim CK, Yi SY, Jang JS, Park K, Kim HJ. Phase II trial of epidermal growth factor ointment for patients with Erlotinib-related skin effects. Support Care Cancer. 2016 Jan;24(1):301-309. doi: 10.1007/s00520-015-2783-9. Epub 2015 Jun 4. PMID 26041481